CLINICAL TRIAL: NCT00026351
Title: Phase II Multicenter Trial Of Pentostatin and Rituximab In Patients With Previously Treated and Untreated Low Grade B-Cell Non-Hodgkin's Lymphoma (NHL) Including Chronic Lymphocytic Leukemia (CLL)
Brief Title: Pentostatin and Rituximab in Treating Patients With Low-Grade Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmatech Oncology (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069021; PHARMATECH-N007; PHARMATECH-20001631; SUPERGEN-PHARMATECH-N007
Record Dates: First submitted 2001-11-09; First posted 2003-06-25 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2002-07

CONDITIONS: Leukemia; Lymphoma
Keywords: stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; prolymphocytic leukemia; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Leukemia, Prolymphocytic; Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab; Pentostatin

INTERVENTIONS:
Biological: rituximab
Drug: pentostatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining chemotherapy with monoclonal antibody therapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining pentostatin and rituximab in treating patients who have non-Hodgkin's lymphoma or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with low-grade B-cell non-Hodgkin's lymphoma or chronic lymphocytic leukemia treated with pentostatin and rituximab.
* Determine the duration of response, median time to progression, and survival of patients treated with this regimen.
* Determine the safety of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive rituximab IV alone on day 1 of course 1 only. Patients then receive rituximab IV and pentostatin IV on days 8, 15, and 22. An additional course with both drugs is administered on days 36, 43, and 50. Patients with progressive disease or a complete response receive no further treatment. Patients with responsive disease, but less than a complete response, receive one additional course of therapy as above.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 50 non-Hodgkin's lymphoma and 50 chronic lymphocytic leukemia patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed low-grade non-Hodgkin's lymphoma

  * REAL classification:

    * B-cell chronic lymphocytic leukemia
    * Prolymphocytic leukemia
    * Small lymphocytic lymphoma
    * Follicular center lymphoma (grade I, II, or III)
    * Extranodal marginal zone B-cell lymphoma Malt type
  * International Working Group classification:

    * Small lymphocytic/chronic lymphocytic leukemia (CLL)

      * CLL with lymph node involvement allowed
    * Small lymphocytic plasmacytoid
    * Follicular small cleaved cell
    * Follicular mixed small and large cell
    * Follicular predominantly large cell
* Measurable disease

  * Lymph node more than 1 cm in longest transverse diameter NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 6 months

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* AST no greater than 5 times upper limit of normal

Renal:

* Creatinine less than 2.0 mg/dL
* BUN normal
* Urinalysis normal

Cardiovascular:

* LVEF normal in patients with history of stable heart disease for at least 2 years

Other:

* HIV negative
* No thyroid disease with thyroid function that cannot be maintained in the normal range
* No other prior malignancy unless progression free for more than 5 years
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior rituximab, Y2B8, or iodine I 131 tositumomab allowed provided at least 6 months have elapsed and patient has had clear disease progression
* No other concurrent immunotherapy

Chemotherapy:

* No more than 6 prior chemotherapy drugs
* No more than 3 prior treatments with pentostatin
* At least 3 weeks since prior chemotherapy
* No prior cumulative lifetime dose of more than 480 mg/m2 of doxorubicin or an equivalent dose of any anthracycline
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No concurrent radiotherapy to an indicator lesion

Surgery:

* Not specified

Other:

* No other concurrent investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Poehlman, Study Chair — Pharmatech Oncology
Locations (5):
- United States (5):
  - Cancer and Blood Institute of the Desert, Rancho Mirage, California
  - Redding Medical Center, Redding, California
  - Oncology-Hematology Associates, P.A., Clinton, Maryland
  - North Shore Hematology/Oncology Associates, P.C., East Setauket, New York
  - Hematology Oncology Associates of Central New York, P.C., Syracuse, New York